CLINICAL TRIAL: NCT05531110
Title: A Randomised, Controlled Study to Compare Visual Performance Following Bilateral, Micro-monovision Insertion of Two Monofocal, Aspheric, Hydrophobic Acrylic Intraocular Lenses: The TECNIS Eyhance® ICB00 and the Alcon IQ SN60WF Lenses
Brief Title: Comparison of Two Aspheric Intraocular Lenses for Micro-monovision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: City, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 315330
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Cataract; Presbyopia; Pseudophakia
Keywords: cataract; pseudophakia; presbyopia
MeSH Terms: conditions — Cataract; Presbyopia; Pseudophakia | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patient will not be informed of which arm of the study they will be allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control arm (Active Comparator): Bilateral Alcon SN60WF IOL insertion
  Interventions: Device: Cataract surgery with insertion of Alcon SN60WF
- Intervention arm (Experimental): Bilateral Eyhance ICB00 IOL
  Interventions: Device: Cataract surgery with insertion of Eyhance ICB00

INTERVENTIONS:
Device: Cataract surgery with insertion of Eyhance ICB00 — Cataract surgery with insertion of Eyhance ICB00
  Arms: Intervention arm
Device: Cataract surgery with insertion of Alcon SN60WF — Cataract surgery with insertion of Alcon SN60WF
  Arms: Control arm

SUMMARY:
In an aging population, cataract and presbyopia become increasingly common. A cataract develops when the natural crystalline lens inside a person's eye, becomes cloudy over time, causing reduction of vision. Presbyopia is an age related condition resulting in loss of reading/near vision and requiring reading glasses.

Cataract surgery is the most common elective surgery in the world for patients over 65. It is composed of removal the cataract and insertion of a new intraocular lens (IOL). Currently only monofocal IOLs are available on the NHS (National Health Service, United Kingdom) - meaning they give good distance or near vision. The majority of patients opt for good distance vision with glasses to read.

The investigators are trialling insertion of a new Extended Depth of Focus (enhanced aspheric) IOL (EDoF IOL), which treats both cataract and presbyopia. All patients attending St Thomas' hospital for treatment of cataracts will be considered for invitation to the study.

Patients who participate in the study will be randomly selected to receive either the new Extended Depth of Focus IOL - the TECNIS Eyhance ICB00 IOL, or a well-established monofocal (non-EDoF) IOL the Alcon Acrysof IQ SN60WF IOL during cataract surgery. Insertion of the Alcon Acrysof IQ SN60WF IOL is known to treat cataract but not presbyopia.

Patients will be assessed and have their surgery performed at St Thomas' Hospital London. They will have 7 appointments over 12 months, plus surgery. The investigators hope to demonstrate better distance, intermediate and near vision and increased spectacle independence in the TECNIS Eyhance ICB00 IOL group.

EDoF IOLs have the potential to improve cataract surgery outcomes for patients in the NHS.

DETAILED DESCRIPTION:
This study is a clinical trial, designed to compare visual outcomes after cataract surgery with two different intraocular lenses. As previously described, modern day cataract surgery is composed of two main components: removal of the cataract, and insertion of an intraocular lens (IOL). The role of the intraocular lens is to replace the focusing power of the natural crystalline lens inside the eye. It is this lens that becomes a cataract. Removing a cataract alone helps light enter the eye, but does not focus it well. Prior to the invention of intraocular lenses, patients required extremely thick and strong glasses for both distance and near vision.

Currently only monofocal intraocular lenses are available on the NHS. Different strengths of lens can be chosen to give the patient good distance, intermediate or near vision. That means the ability to focus on objects in the distance, middle distance or near. Most patients opt for good distance vision, enabling them to mobilise easily, watch TV and drive, and require glasses for reading.

As described above, most patients over the age of 50, have some element of presbyopia, which is the inability to focus on near objects, resulting in the need for reading glasses. Inserting extended depth of focus (EDoF IOLs) intraocular lenses during cataract surgery, can help improve their reading vision without reading glasses.

The TECNIS Eyhance ICB00 IOL is a new EDoF IOL which has an enhanced depth of focus through its novel 'enhanced aspheric' design. This will help treat presbyopia. The Alcon Acrysof IQ SN60WF IOL is an established IOL which gives good monofocal vision, i.e. good distance or near vision, but not both.

Our trial will investigate the effect of a new Extended depth of focus lens on vision and compare it to a commonly used Monofocal IOL. The investigators will recruit patients who have bilateral cataracts. These patients will have otherwise healthy eyes. Patients who have been referred to St Thomas' Hospital for assessment for cataracts will be considered for the trial. If they fulfil the criteria for acceptance to the trial, the consulting doctor will discuss this with the patient. If the patient expresses interest, they will be referred to the Research department. The cataract research fellow will review them and consider them for admission to the trial. This review will happen on the day of the original appointment, or the patient will be given an another appointment time and date for further assessment. If a patient would like further information about the study, but cannot speak to the Cataract Research Fellow that same day, they will be asked to fill in a Consent to Contact form, which will allow the research department to contact the patient for consideration for entry to the study.

The investigators will recruit 2 groups of patients, with 70 patients in each group. The investigators will randomly assign them to either the TECNIS Eyhance ICB00 group or the Alcon Acrysof IQ SN60WF IOL group. Patients will not be informed of which group they are in, until completion of the study. This 'masking' is to help reduce bias in the post-operative testing. Although the Doctors in the research dept will know which group the patient is in, by not giving this information to the patient, the investigators aim to get a more accurate assessment of their satisfaction with their vision.

All patients will have cataract surgery on one eye, an appointment to review their post-operative outcome, and then the second cataract operation. The patients in the TECNIS Eyhance group will have TECNIS Eyhance ICB00 lenses inserted into both eyes. The patients in the Alcon group will have Alcon Acrysof IQ SN60WF lenses inserted into both eyes. Patients who fulfil the inclusion/exclusion criteria will be fully informed of the investigative nature of the study and consented. The TECNIS Eyhance ICB00 IOL is not used in the NHS, but is used in private practice in the UK. The Alcon SN60WF IOL is commonly used in the NHS.

Once patients are consented, they will have a standard pre-operative assessment which will include taking a medical and ophthalmic history, a full eye examination, refraction (similar to an assessment with an optician), have their vision tested at distance with and without glasses, and an intraocular pressure check (tonometry). The investigators will perform a biometry (measurement of the eye) to calculate the lens power required for surgery. Intraocular lenses are available in different powers, in the same way spectacle lenses are available in different powers. The investigators will also document the type of glasses a patient uses. The investigators will also perform a Macula OCT scan - a non invasive scan of the macula, which is the central part of the retina. The investigators will also perform an endothelial cell count, which is an non-invasive scan of the inner layer fo the cornea.

Cataract surgery will be performed during NHS cataract lists at St Thomas' Hospital. Surgery will be performed by senior cataract surgeons, and standard protocols will be followed. The investigators will endevour to reduce astigmatism using on-axis incisions and opposite clear corneal incisions (OCCIs). These are standard cataract surgery techniques.

The investigators will be using a strategy called micro-monovision. Most people have a dominant eye, in the same way that they have a dominant hand. In micro-monovision the investigators choose an intraocular lens power that will give the dominant eye good distance vision (emmetropia), and a intraocular lens power that will give the non-dominant eye good intermediate distance vision. The investigators will be using this strategy in both the TECNIS Eyhance ICB00 group and the Alcon IQ SN60WF group.

Post-operatively patients will be processed in the usual manner based on the protocol developed for cataract surgery at our institution (Guy's and St. Thomas' NHS Foundation Trust, London, UK) and will undergo an out-patient appointment 2 weeks.

During this appointment the investigators will assess the patient's vision (unaided, with glasses and with pinhole), intraocular pressure (tonometry), refraction (with an autorefraction machine), perform a full eye examination, included dilation of the pupils and fundoscopy. The investigators will also perform a macula OCT scan.

As well as the standard and pre- and post operative assessments, patients will have the following additional Appointments and investigations

Patients will be asked to return at 6 weeks and 6 months after each eye operation, a total 4 extra appointments. In addition to the standard tests performed as part of pre- and post-operative assessment for cataract surgery the investigators will perform the following tests.

Visual acuity testing:

It is standard to record near and distance vision before and after cataract surgery. The investigators will also assess middle-distance vision at 66 cm. The investigators will assess this at all appointments.

Slit lamp biomicroscopy, tonometry & dilated funduscopy:

At 6 weeks and 6-months following each eye surgery patients will be asked to attend out-patient visits during which they will have slit lamp examination, tonometry and dilated fundoscopy, as they have had done at enrolment.

A slit lamp is the microscope that an ophthalmologist or optician uses to examine the eye. Patients will have dilating drops applied to each eye (described below). These cause temporary dilation of the pupils which allow examination of the back of the eye, called dilated fundoscopy. Tonometry refers to measurement of the pressure of the eye.

Endothelial Cell Count This is an automated non-contact, non-invasive, specular microscope which produces and image and cell count of the inner layer of the cornea. It will be performed at preassessment, as well as 6 weeks and 6 months after each eye operation.

Dilating Eyedrops:

1 drop of each of 1% Tropicamide, and 2.5% phenylephrine will be instilled to each eye at every appointment to allow for complete examination of the eye.

Glasses:

At enrolment, the investigators will gather information on what glasses they currently use. The investigators will then ask them again at 6 months after each eye operation, and compare this with pre-operative data.

Contrast sensitivity:

The investigators will assess contrast sensitivity of both eyes at enrolment, and then the contrast sensitivity of the operated eye, 6 weeks & 6 months after each operation.

Stereoacuity:

The investigators will assess stereoacuity at enrolment and then 6 weeks and 6 months after the second eye operation.

Refraction:

The investigators will perform autorefraction at enrolment, 2 weeks, 6 weeks, and 6 months after surgery. The investigators will perform subjective refraction at 6 weeks and 6 months after surgery.

Refraction is a measurement of a patient's refractive error. This is measured in dioptres, and is used to generate a glasses prescription. Autorefraction refers to an automated measurement performed by a machine called an autorefractor. Subjective refraction is performed by an optometrist or ophthalmologist.

Schiempflug tomography/topography (Pentacam):

The investigators will perform this at enrolment, 6 weeks and 6 months after eye surgery. This will be performed to assess IOL decentration and tilt.

Macula OCT:

This is routinely performed before and after cataract surgery, to exclude cystoid macula oedema. The investigators will perform this as well at 6 weeks and 6 months after surgery.

Digital photograpy:

After instillation of dilating eyedrops, the investigators will perform intraocular lens photography to assess capsular opacification and lens glistenings at 6 months after surgery in either eye. Anonymised digital images may be shared with Prof Chris Hull at City University to help us assess glistening of the IOLs.

Questionnaires:

At enrolment, 6 weeks and 6-months visits, patients will be asked to complete PROM questionnaires, namely EQ-5D-3L, Catquest and Cat-PROM5. These questionnaires assess a patient's general health and attitudes to their vision.

Adverse events:

The investigators will document any adverse events at every appointment.

The investigators estimate it will take patients 120 minutes to complete this study enrolment / consent and extra investigations

Interim data will be reviewed at 20% completion of treatment and 6 month followup (following second eye surgery). The study completion date will be when Patient 140 has completed their 6 month visit (following second eye surgery) plus 14 days for data entry and database lock.

The investigators are testing the following hypotheses (theories)

1. That bilateral, micro-monovision TECNIS Eyhance® ICB00 IOL implantation will achieve superior intermediate and near unaided visual performance compared to bilateral, micro-monovision implantation of the Alcon IQ SN60WF lens, while maintaining similar distance vision performance, contrast sensitivity and dysphotopsia occurrences.
2. That bilateral, micro-monovision TECNIS Eyhance® ICB00 IOL implantation will achieve higher patient satisfaction (PROMs) scores due to superior intermediate, and near unaided visual performance compared to bilateral, micro-monovision implantation of the Alcon IQ SN60WF monofocal IOL.
3. That bilateral, micro-monovision TECNIS Eyhance® ICB00 IOL implantation will be more cost effective in terms of patient expenditure on intermediate and complex (bifocals, varifocals) near vision spectacles due to superior intermediate, and near unaided visual performance compared to bilateral, micro-monovision implantation of standard aspheric monofocal IOLs.

ELIGIBILITY:
Inclusion Criteria:

- Bilateral cataract requiring surgical intervention, age over 18 years able to understand informed consent and the objectives of the trial, not pregnant, not breast feeding no previous intraocular eye surgery good visual potential in both eyes corneal astigmatism of less than 1.5 diopters

Exclusion Criteria:

-

Any patient with other ocular condition that might reduce visual acuity and hence confound the results such as:

1. visually impairing age-related macular degeneration
2. Advanced glaucoma
3. previous retinal vascular disorders
4. previous retinal detachment or tear
5. any visually impairing neuro-ophthalmological condition
6. any inherited retinal disorder or pathology
7. previous strabismus surgery or record of amblyopia
8. previous visually impairing CVA, TIA or other vaso-occlusive disease
9. already enrolled in another study or trial
10. instability of keratometry or biometry measurements
11. irregular astigmatism
12. previous significant trauma to eye
13. age over 100

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Acuity from baseline to 6 weeks | 6 weeks after cataract surgery
  Uniocular & Binocular, Unaided and Best Corrected, Near, intermediate and distance vision
Change in Visual Acuity from baseline to 6 months | 6 months after cataract surgery
  Uniocular & Binocular, Unaided and Best Corrected, Near, intermediate and distance vision
Change in Refractive Error from baseline to 6 weeks | 6 weeks after cataract surgery
  Optometrist assessed refractive error for Near, and distance vision
Change in Refractive Error from baseline to 6 months | 6 months after cataract surgery
  Optometrist assessed refractive error for Near, and distance vision
Change in Patient Satisfaction from baseline to 6 weeks | baseline and 6 weeks after cataract surgery
  Patient satisfaction - PROM questionnaire: EQ-5D-3L scores A 2 part questionnaire
  1. 5 questions, with 3 options each. Each question is scored 1 to 3, with the cumulative assessment described as a 5 digit code.
  2. The second part asks patients to estimate their health on the day of the questionnaire on a numerical and visual scale ranging from 0 (worst health possible) to 100 (best health imaginable).
Change in Patient Satisfaction from baseline to 6 weeks | baseline and 6 weeks after cataract surgery
  patient satisfaction - PROM questionnaire: Catquest-9SF scores 9 item questionnaire with 4 options each, can be converted to a numerical score (9-36), with 36 being the worst vision
Change in Patient Satisfaction from baseline to 6 weeks | baseline and 6 weeks after cataract surgery
  patient satisfaction - PROM questionnaire: Cat-PROM scores 5 question questionnaire which gives a converted Rasch score, from 0-100, with 100 the best vision
Change in Patient Satisfaction from baseline to 6 months | baseline and 6 months after cataract surgery
  patient satisfaction - PROM questionnaire: EQ-5D-3L scores
  A 2 part questionnaire
  1. 5 questions, with 3 options each. Each question is scored 1 to 3, with the cumulative assessment described as a 5 digit code.
  2. The second part asks patients to estimate their health on the day of the questionnaire on a numerical and visual scale ranging from 0 (worst health possible) to 100 (best health imaginable).
Change in Patient Satisfaction from baseline to 6 months | baseline and 6 months after cataract surgery
  Patient satisfaction - PROM questionnaire: Catquest-9SF scores 9 item questionnaire with 4 options each, can be converted to a numerical score (9-36), with 36 being the worst vision
Change in Patient Satisfaction from baseline to 6 months | baseline and 6 months after cataract surgery
  PROM questionnaire : Cat-PROM scores 5 question questionnaire which gives a converted Rasch score, from 0-100, with 100 the best vision
Change in Cost Benefits from baseline to 6 weeks | 6 weeks after cataract surgery
  Patient related cost benefits in terms of spectacle expenditure.
Change in Cost Benefits from baseline to 6 months | 6 months after cataract surgery
  Patient related cost benefits in terms of spectacle expenditure.

SECONDARY OUTCOMES:
Change in Contrast Sensitivity at 6 weeks after surgery | 6 weeks after cataract surgery
  CVS-1000
Change in Contrast Sensitivity at 6 months after surgery | 6 months after cataract surgery
  CVS-1000
Change in Stereoacuity at 6 weeks after cataract surgery | 6 weeks after the second cataract surgery
  Randot test
Change in Stereoacuity at 6 months after cataract surgery | 6 months after the second cataract surgery
  Randot
Documentation of Post-operative complications 2 weeks after surgery | 2 weeks after cataract surgery
  Documentation of post-operative complications including: IOL decentration, tilt, posterior capsule Opacification, dysphotopsias
Documentation of Post-operative complications 6 weeks after surgery | 6 weeks after cataract surgery
  Documentation of post-operative complications including: IOL decentration, tilt, posterior capsule Opacification, dysphotopsias
Documentation of Post-operative complications | 6 months after cataract surgery
  Documentation of post-operative complications including: IOL decentration, tilt, posterior capsule Opacification, dysphotopsias

CONTACTS AND LOCATIONS:
Overall Officials: David O'Brart, MBBS, MD, Study Director — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No